CLINICAL TRIAL: NCT01121393
Title: LUX-Lung 6: A Randomized, Open-label, Phase III Study of BIBW 2992 Versus Chemotherapy as First-line Treatment for Patients With Stage IIIB or IV Adenocarcinoma of the Lung Harbouring an EGFR Activating Mutation
Brief Title: BIBW 2992 (Afatinib) vs Gemcitabine-cisplatin in 1st Line Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1200.34
Record Dates: First submitted 2010-04-21; First posted 2010-05-12 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Adenocarcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Adenocarcinoma | interventions — Afatinib

ARMS (2):
- Arm A BIBW 2992 (Experimental): Patients receive a tablet of BIBW 2992 daily until progression or unacceptable toxicity
  Interventions: Drug: BIBW 2992
- Arm B Chemotherapy (Active Comparator): Patients receive Gemcitabine and Cisplatin, maximum is 6 courses
  Interventions: Drug: Gemcitabine+Cisplatin

INTERVENTIONS:
Drug: Gemcitabine+Cisplatin — Gemcitabine d1,8, Cisplatin d1, 21 days as a course, up to 6 courses.
  Arms: Arm B Chemotherapy
Drug: BIBW 2992 — starting dose is 40 mg, in the event of no or minimal drug-related adverse events after one course, the dose will be increased to 50mg. in the event of certain drug related Adverse Event (AE), dose reduction will be increments of 10 mg, with the lowest dose being 20mg.
  Arms: Arm A BIBW 2992

SUMMARY:
To investigate the efficacy and safety of BIBW 2992 compared to standard first-line chemotherapy in patients with stage IIIB or IV adenocarcinoma of the lung harbouring an EGFR activating mutation

ELIGIBILITY:
Inclusion criteria:

1. pathologically confirmed diagnosis of stage IIIB or stage IV adenocarcinoma of the Lung
2. EGFR(Epidermal Growth Factor Receptor) mutation detected by central laboratory analysis of tumor biopsy material
3. Measurable disease according to Response Evaluation Criteria in Solid Tumours (RECIST)1.1
4. Eastern Cooperative Oncology Group (ECOG) score of 0 or 1.
5. Age>=18 years
6. life expectancy of at least three months
7. Written informed consent that is consistent with International Conference on Harmonisation-Good Clinical Practice (ICH-GCP) guidelines.

Exclusion criteria:

1. Prior chemotherapy for relapsed and/or metastatic NSCLC.
2. Prior treatment with EGFR targeting small molecules or antibodies.
3. Radiotherapy or surgery(other than biopsy) within 4 weeks prior to randomization
4. Active brain metastases
5. Any other current malignancy or malignancy diagnosed within the past 5 years
6. Known pre-existing interstitial lung disease
7. Significant or recent acute gastrointestinal disorders with diarrhoea as a a major symptoms.
8. History or presence of clinically relevant cardiovascular abnormalities
9. Cardiac left ventricular function with resting ejection fraction of less than 50%.
10. Any other concomitant serious illness or organ system dysfunction which in the opinion of the investigator would either compromise patient safety or interfere with the evaluation of the safety of the test drug.
11. Absolute neutrophil count(ANC)<1500/mm3
12. Platelet count<100,000/mm3
13. Creatinine clearance<60ml/min or serum creatinine>1.5 times Upper Limit of Normal (ULN).
14. Bilirubin>1.5 times ULN
15. Aspartate Amino Transferase (AST) or Alanine Amino Transferase (ALT) > 3 times ULN
16. Women of childbearing potential, or men who are able to father a child, unwilling to use a medically acceptable method of contraception during the trial
17. Pregnancy of breast-feeding
18. Patients unable to comply with the protocol
19. Active hepatitis B infection, active hepatitis C infection or known HIV(Human Immunodeficiency Virus) carrier.
20. Known or suspected active drug or alcohol abuse.
21. requirement for treatment with any of the prohibited concomitant medications listed in section 4.2.2
22. Any contraindications for therapy with gemcitabine/cisplatin
23. Known hypersensitivity to BIBW2992 or the excipient of any of the trial drugs
24. Use of any investigational drug within 4 weeks of randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Actual)
Dates: Start 2010-04-19 (Actual); Primary Completion 2017-11-23 (Actual); Study Completion 2017-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (36):
- China (30):
  - Beijing Chao-Yang Hospital, Beijing
  - 307 Hospital of PLA, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Beijing Chest Hospital, Beijing
  - First Hospital of Jilin University, Changchun
  - Xiangya Hospital, Central South University, Changsha
  - Hunan Province Tumor Hospital, Changsha
  - West China Hospital, Chengdu
  - Fujian Provincial Tumor Hospital, Fuzhou
  - Guangdong General Hospital, Guangzhou
  - Guangzhou Institute of Respiratory Disease, Guangzhou
  - NanFang Hosptial, Guangzhou
  - The Third Affiliated Hospital of Harbin Medical University, Haerbin
  - Zhejiang Cancer Hospital, Hangzhou
  - Hubei Cancer Hospital, Hongshan
  - Yunnan Provincial Tumor Hospital, Kunming
  - Lin Yi Tumor Hospital, Linyi
  - the 81th Hospital of PLA, Nanjing
  - Jiangsu Cancer Hospital, Nanjing
  - The Affiliated Cancer Hospital, Guangxi Medical University, Nanning
  - The affiliated hospital of medicalcollege qingdao university, Qingdao
  - Shanghai Changzheng Hospital, Shanghai
  - Shanghai Chest Hospital, Shanghai
  - Zhongshan Hospital Fudan University, Shanghai
  - Shanghai Pulmonary Hospital, Shanghai
  - Changhai Hospital, Shanghai
  - The First Hospital of Chinese Medical University, Shenyang
  - Hebei Provincial Tumor Hospital, Shijiazhuang
  - Tangdu Hospital, Xi'an
  - Northern Jiangsu People's Hospital, Yangzhou
- South Korea (5):
  - Kosin University Gospel Hospital, Busan
  - Chungbuk National University Hospital, Cheongju-si
  - Yeungnam University Medical Center, Daegu
  - Konkuk University Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
- Songklanagarind Hospital, Songkhla, Thailand

REFERENCES:
- [Derived] Wu YL, Xu CR, Hu CP, Feng J, Lu S, Huang Y, Li W, Hou M, Shi JH, Marten A, Fan J, Peil B, Zhou C. Afatinib versus gemcitabine/cisplatin for first-line treatment of Chinese patients with advanced non-small-cell lung cancer harboring EGFR mutations: subgroup analysis of the LUX-Lung 6 trial. Onco Targets Ther. 2018 Nov 30;11:8575-8587. doi: 10.2147/OTT.S160358. eCollection 2018. PMID 30584317
- [Derived] Wu YL, Sequist LV, Tan EH, Geater SL, Orlov S, Zhang L, Lee KH, Tsai CM, Kato T, Barrios CH, Schuler M, Hirsh V, Yamamoto N, O'Byrne K, Boyer M, Mok T, Peil B, Marten A, Chih-Hsin Yang J, Paz-Ares L, Park K. Afatinib as First-line Treatment of Older Patients With EGFR Mutation-Positive Non-Small-Cell Lung Cancer: Subgroup Analyses of the LUX-Lung 3, LUX-Lung 6, and LUX-Lung 7 Trials. Clin Lung Cancer. 2018 Jul;19(4):e465-e479. doi: 10.1016/j.cllc.2018.03.009. Epub 2018 Mar 17. PMID 29653820
- [Derived] Yang JC, Sequist LV, Zhou C, Schuler M, Geater SL, Mok T, Hu CP, Yamamoto N, Feng J, O'Byrne K, Lu S, Hirsh V, Huang Y, Sebastian M, Okamoto I, Dickgreber N, Shah R, Marten A, Massey D, Wind S, Wu YL. Effect of dose adjustment on the safety and efficacy of afatinib for EGFR mutation-positive lung adenocarcinoma: post hoc analyses of the randomized LUX-Lung 3 and 6 trials. Ann Oncol. 2016 Nov;27(11):2103-2110. doi: 10.1093/annonc/mdw322. Epub 2016 Sep 6. PMID 27601237
- [Derived] Schuler M, Wu YL, Hirsh V, O'Byrne K, Yamamoto N, Mok T, Popat S, Sequist LV, Massey D, Zazulina V, Yang JC. First-Line Afatinib versus Chemotherapy in Patients with Non-Small Cell Lung Cancer and Common Epidermal Growth Factor Receptor Gene Mutations and Brain Metastases. J Thorac Oncol. 2016 Mar;11(3):380-90. doi: 10.1016/j.jtho.2015.11.014. Epub 2016 Jan 25. PMID 26823294
- [Derived] Yang JC, Sequist LV, Geater SL, Tsai CM, Mok TS, Schuler M, Yamamoto N, Yu CJ, Ou SH, Zhou C, Massey D, Zazulina V, Wu YL. Clinical activity of afatinib in patients with advanced non-small-cell lung cancer harbouring uncommon EGFR mutations: a combined post-hoc analysis of LUX-Lung 2, LUX-Lung 3, and LUX-Lung 6. Lancet Oncol. 2015 Jul;16(7):830-8. doi: 10.1016/S1470-2045(15)00026-1. Epub 2015 Jun 4. PMID 26051236
- [Derived] Yang JC, Wu YL, Schuler M, Sebastian M, Popat S, Yamamoto N, Zhou C, Hu CP, O'Byrne K, Feng J, Lu S, Huang Y, Geater SL, Lee KY, Tsai CM, Gorbunova V, Hirsh V, Bennouna J, Orlov S, Mok T, Boyer M, Su WC, Lee KH, Kato T, Massey D, Shahidi M, Zazulina V, Sequist LV. Afatinib versus cisplatin-based chemotherapy for EGFR mutation-positive lung adenocarcinoma (LUX-Lung 3 and LUX-Lung 6): analysis of overall survival data from two randomised, phase 3 trials. Lancet Oncol. 2015 Feb;16(2):141-51. doi: 10.1016/S1470-2045(14)71173-8. Epub 2015 Jan 12. PMID 25589191
- [Derived] Wu YL, Zhou C, Hu CP, Feng J, Lu S, Huang Y, Li W, Hou M, Shi JH, Lee KY, Xu CR, Massey D, Kim M, Shi Y, Geater SL. Afatinib versus cisplatin plus gemcitabine for first-line treatment of Asian patients with advanced non-small-cell lung cancer harbouring EGFR mutations (LUX-Lung 6): an open-label, randomised phase 3 trial. Lancet Oncol. 2014 Feb;15(2):213-22. doi: 10.1016/S1470-2045(13)70604-1. Epub 2014 Jan 15. PMID 24439929

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two-arm, randomised (2:1 ratio), open-label, active-controlled, parallel-group comparison of afatinib versus gemcitabine / cisplatin chemotherapy.
Pre-assignment Details: All patients were screened for eligibility to participate in the trial. Patients attended a specialist sites which ensured that they met all strictly implemented inclusion/exclusion criteria. Patients were not to be entered to trial treatment if any one of the specific entry criteria was violated.
Groups:
- Afatinib 40 Milligram (mg): Patients received Afatinib film-coated tablets 40 mg once daily (q.d.) orally with possible dose escalation to 50 mg q.d. and dose reduction to 40 mg q.d. (if applicable), 30 mg q.d., or 20 mg q.d. (according to the protocol-defined dose-escalation and dose-reduction scheme), if required. No dose increase was allowed after dose reduction. Each treatment course was planned to be 21 days. For afatinib, patients received continuous daily dosing until disease progression, unacceptable adverse events (AEs) occurred, or withdrawal of consent for any reason.
- Gemcitabine / Cisplatin Chemotherapy: Patients received Gemcitabine (lyophilised powder) 1000 milligram per square metre (mg/m²) as an intravenous infusion over 30 minutes on day 1 and day 8, cisplatin (solution for infusion) 75 mg/m² as an intravenous infusion on Day 1 of each 21-day treatment course up to 6 cycles; Chemotherapy could be delayed or the dose could be reduced in accordance with the guidance in the current summary of product characteristics. For gemcitabine / cisplatin, patients were to receive a maximum of 6 treatment courses unless they developed disease progression, experienced unacceptable AEs, or withdrawal of consent for any reason.
Period: Overall Study
Arm/Group | Afatinib 40 Milligram (mg) | Gemcitabine / Cisplatin Chemotherapy
Started | 242 (Randomised) | 122 (Randomised)
Treated | 239 (Treated) | 113 (Treated)
Completed | 0 (At the time of data cut-off for last-patient out (07 December 2017)) | 38 (Completed 6 courses of chemotherapy)
Not Completed | 242 | 84
Not completed — Progressive disease | 201 | 20
Not completed — Other Adverse events | 24 | 45
Not completed — Non-compliant with protocol | 0 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Refused cont. medication | 7 | 7
Not completed — Not treated | 3 | 9
Not completed — Other than listed | 6 | 0

BASELINE CHARACTERISTICS:
Population: The randomised set (RS) included all patients randomised to receive treatment, whether treated or not.
Groups:
- Total: Total of all reporting groups
Arm/Group | Afatinib 40 Milligram (mg) | Gemcitabine / Cisplatin Chemotherapy | Total
Number analyzed (Participants) | 242 | 122 | 364
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Treated Set
  Years | 56.7 (11.2) | 55.6 (10.1) | 56.4 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 155 | 83 | 238
  Male | 87 | 39 | 126
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Epidermal growth factor receptor (EGFR) [Count of Participants; unit: Participants] — EGFR mutation group (L858R / Deletion Exon 19 / other) was a stratification factor.
  Participants
    L858R (L858R alone and L858R + Deletion Exon 19) | 92 | 46 | 138
    Deletion Exon 19 (alone) | 124 | 62 | 186
    Other | 26 | 14 | 40
Eastern Cooperative Oncology Group (ECOG) performance status (PS) [Count of Participants; unit: Participants] — ECOG PS measured on 6 point scale to assess participant's performance status. 0=Fully active, able to carry on all pre-disease activities without restriction; 1=Restricted in physically strenuous activity, but ambulatory and able to carry out light or sedentary work; 2=Ambulatory (>50 percent of waking hours), capable of all selfcare, unable to carry out any work activities; 3=Capable of only limited self care, confined to bed or chair more then 50 percent of waking hours; 4=Completely disabled, cannot carry on any selfcare, totally confined to bed or chair; 5=Dead
  Participants
    ECOG PS 0 (baseline) | 48 | 41 | 89
    ECOG PS 1 (baseline) | 194 | 81 | 275

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: The primary endpoint was progression-free survival (PFS) as assessed by central independent review according to Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1. Progression-free survival was defined as the time from randomisation to disease progression or death whichever occurs earlier. A pre-defined set of censoring rules were used for patients who did not have a PFS.
  Only data collected up until the analysis cut-off date (27 December 2013) were considered. Median time results from unstratified Kaplan-Meier estimates.
Time Frame: Tumour assessment were performed at screening, week 6, 12, 18, 24, 30, 36, 42, 48 and then every 12 weeks until progression or death whichever occurs first up to week 168
Population: The randomised set (RS) included all patients randomised to receive treatment, whether treated or not.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Afatinib 40 Milligram (mg) | Gemcitabine / Cisplatin Chemotherapy
Number analyzed (Participants) | 242 | 122
months | 11.01 [9.66 to 13.73] | 5.59 [4.67 to 6.70]
Statistical Analysis 1: Comparison: Afatinib 40 Milligram (mg) vs Gemcitabine / Cisplatin Chemotherapy; A stratified log-rank test (by the epidermal growth factor receptor (EGFR) mutation category stratification factor used at randomisation) was used to test for the effect of afatinib on PFS compared with gemcitabine / cisplatin chemotherapy; Test type: Superiority; p < 0.0001, Log Rank
Statistical Analysis 2: Comparison: Afatinib 40 Milligram (mg) vs Gemcitabine / Cisplatin Chemotherapy; A Cox proportional-hazards model, stratified by EGFR mutation category was used to estimate the hazard ratio (HR) and 95% confidence interval (CI) between the 2 treatment arms; Test type: Superiority; Hazard Ratio (HR) = 0.281, 95% CI 2-sided [0.203 to 0.389]

2. Secondary Outcome: Objective Response (OR)
Description: OR is defined as a best overall response of complete response (CR) or partial response (PR) assessed by central independent review according to RECIST version 1.1 and will be presented as the percentage of patients with OR.
  CR is defined as the disappearance of all target lesions and non-target lesions and no new lesions.
  PR is defined as at least a 30% decrease in the sum of longest diameter (LD) of target lesions taking as reference the baseline sum LD, non-Progressive Disease or non evaluation of all non-target lesions and no new lesions.
  (Exact 95% Confidence interval by Clopper and Pearson.)
Time Frame: Tumour assessment were performed at screening, week 6, 12, 18, 24, 30, 36, 42, 48 and then every 12 weeks until progression or death whichever occurs first up to week 374
Population: The randomised set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Afatinib 40 Milligram (mg) | Gemcitabine / Cisplatin Chemotherapy
Number analyzed (Participants) | 242 | 122
percentage of participants | 67.8 [61.5 to 73.6] | 23.0 [15.8 to 31.4]
Statistical Analysis 1: Comparison: Afatinib 40 Milligram (mg) vs Gemcitabine / Cisplatin Chemotherapy; A logistic regression model, stratified by EGFR mutation category was used to compare the objective response rate between the 2 treatment arms; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 7.572, 95% CI 2-sided [4.522 to 12.679]

3. Secondary Outcome: Disease Control (DC)
Description: DC is defined as a patient with objective response (OR) or stable disease (SD) assessed by central independent review according to RECIST version 1.1 and will be presented as the percentage of patients with DC.
Time Frame: as for outcome 2
Population: The randomised set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Afatinib 40 Milligram (mg) | Gemcitabine / Cisplatin Chemotherapy
Number analyzed (Participants) | 242 | 122
percentage of participants | 92.6 [88.5 to 95.5] | 76.2 [67.7 to 83.5]
Statistical Analysis 1: Comparison: Afatinib 40 Milligram (mg) vs Gemcitabine / Cisplatin Chemotherapy; stratified for EGFR mutation group; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 3.843, 95% CI 2-sided [2.039 to 7.240]

4. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from randomisation to death. For patients who had not died until 7 December 2017, the date they were last known to be alive was derived from patient status records, the trial completion record, radiological imaging assessments, the study treatment termination record, and the randomisation date.
  Median time results from unstratified Kaplan-Meier estimates.
Time Frame: From randomisation up to 374 weeks
Population: The randomised set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Afatinib 40 Milligram (mg) | Gemcitabine / Cisplatin Chemotherapy
Number analyzed (Participants) | 242 | 122
months | 23.10 [20.40 to 27.33] | 23.46 [17.94 to 25.56]
Statistical Analysis 1: Comparison: Afatinib 40 Milligram (mg) vs Gemcitabine / Cisplatin Chemotherapy; A stratified log-rank test (by the epidermal growth factor receptor (EGFR) mutation category stratification factor used at randomisation) was used to test for the effect of afatinib on OS compared with gemcitabine / cisplatin chemotherapy; Test type: Superiority; p = 0.4013, Log Rank
Statistical Analysis 2: Comparison: Afatinib 40 Milligram (mg) vs Gemcitabine / Cisplatin Chemotherapy; A Cox proportional hazard model stratified (by EGFR mutation category stratification factor used at randomisation) was used to test the effect of afatinib on OS compared with gemcitabine / cisplatin chemotherapy; Test type: Superiority; Hazard Ratio (HR) = 0.904, 95% CI 2-sided [0.715 to 1.144]

5. Secondary Outcome: Time to Objective Response (OR)
Description: OR is defined as a best of overall response of complete response (CR) or partial response (PR) assessed by central independent review according to RECIST version 1.1.
  For patients with an objective response, time to objective response was defined as the time from randomisation to the first objective response.
  Outcome data are the percentage of patients with OR by each scheduled tumour assessment.
Time Frame: as for outcome 2
Population: The RS included all patients randomised to receive treatment, whether treated or not.
Measure: Number; unit: percentage of participants
Arm/Group | Afatinib 40 Milligram (mg) | Gemcitabine / Cisplatin Chemotherapy
Number analyzed (Participants) | 242 | 122
percentage of participants
  By Week 6 | 49.2 | 13.1
  By Week 12 | 59.9 | 19.7
  By Week 18 | 64.0 | 23.0
  By Week 24 | 64.9 | 23.0
  By Week 30 | 65.7 | 23.0
  By Week 36 | 66.1 | 23.0
  By Week 42 | 66.5 | 23.0
  By Week 48 | 66.5 | 23.0
  By Week 60 | 66.9 | 23.0
  By Week 72 | 66.9 | 23.0
  By Week 84 | 66.9 | 23.0
  By Week 96 | 67.4 | 23.0
  By Week 108 | 67.4 | 23.0
  By Week 120 | 67.8 | 23.0

6. Secondary Outcome: Duration of Objective Response
Description: OR is defined as a best of overall response of complete response (CR) or partial response (PR) assessed by central independent review according to RECIST version 1.1.
  For patients with an objective response, duration of objective response was defined as the time from the first objective response to disease progression or death whichever occurs earlier. A pre-defined set of censoring rules were used for patients who did not progress/die. The Median values are Kaplan-Meier estimates.
Time Frame: as for outcome 2
Population: The Randomised set with an objective response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Afatinib 40 Milligram (mg) | Gemcitabine / Cisplatin Chemotherapy
Number analyzed (Participants) | 164 | 28
months | 9.72 [8.34 to 12.45] | 4.27 [2.76 to 5.75]

7. Secondary Outcome: Duration of Disease Control
Description: For patients with disease control, duration of disease control was defined as the time from randomisation to progression or death whichever occurs first. A pre-defined set of censoring rules were used for patients who did not progress/die. The Median values are Kaplan-Meier estimates.
Time Frame: as for outcome 2
Population: The randomised set with disease control.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Afatinib 40 Milligram (mg) | Gemcitabine / Cisplatin Chemotherapy
Number analyzed (Participants) | 224 | 93
months | 11.07 [9.69 to 13.80] | 5.65 [5.49 to 6.93]

8. Secondary Outcome: Tumour Shrinkage
Description: Tumour shrinkage is calculated as the minimum post-baseline sum of longest diameters of target lesions (longest for non-nodal lesions, short axis for nodal lesions) (SLD), as assessed by central independent review. The mean of these minimum values are presented after adjusting for baseline sum of longest diameters and EGFR mutation category. Only data collected up until the analysis cut-off date (27 Dec 2013) were considered. A negative value means the smallest post-baseline SLD was smaller than baseline (decreased since baseline); a positive value means tumor size increased since baseline.
  The means are adjusted for baseline sum of lesions and EGFR mutation category.
Time Frame: as for outcome 2
Population: The randomised set. There were ony 220 patients in the Afatinib arm and 101 patients in the Gemcitabine / Cisplatin arm with baseline and post-baseline target lesion measurements.
Measure: Mean (Standard Error); unit: millimetre (mm)
Arm/Group | Afatinib 40 Milligram (mg) | Gemcitabine / Cisplatin Chemotherapy
Number analyzed (Participants) | 220 | 101
millimetre (mm) | 33.41 (0.99) | 47.06 (1.45)
Statistical Analysis 1: Comparison: Afatinib 40 Milligram (mg) vs Gemcitabine / Cisplatin Chemotherapy; Test type: Superiority; p < 0.0001, ANCOVA; adjusted for baseline sum of diameters and EGFR mutation group; Mean Difference (Final Values) = -13.64, 95% CI 2-sided [-17.10 to -10.19], Standard Error of Mean 1.76

9. Secondary Outcome: Change From Baseline in Body Weight
Description: The change from baseline to the lowest and the last body weight recorded or during the the study.
Time Frame: Baseline and throughout the study (every 3 weeks) until progression or death (whichever occurs first) up to 374 weeks.
Population: The randomised set. Data only presented for a patient with a baseline and at least on post-baseline assessment of weight.
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | Afatinib 40 Milligram (mg) | Gemcitabine / Cisplatin Chemotherapy
Number analyzed (Participants) | 237 | 109
kilogram (kg)
  Change from baseline at lowest value | -3.03 (3.99) | -1.52 (3.65)
  Change from baseline at last value | -0.76 (4.79) | 0.00 (4.52)

10. Secondary Outcome: Change From Baseline in Eastern Cooperative Oncology Group (ECOG) Performance Status (PS)
Description: The last ECOG performance score category recorded during the study. Outcome data are the percentage of patients with an shift of ECOG performance status from baseline to the last ECOG performance status.
  ECOG PS measured on 6 point scale to assess participant's performance status. 0=Fully active, able to carry on all pre-disease activities without restriction;
  1. Restricted in physically strenuous activity, but ambulatory and able to carry out light or sedentary work;
  2. Ambulatory (>50 percent of waking hours), capable of all selfcare, unable to carry out any work activities;
  3. Capable of only limited self care, confined to bed or chair more then 50 percent of waking hours;
  4. Completely disabled, cannot carry on any selfcare, totally confined to bed or chair;
  5. Dead
Time Frame: Baseline and throughout the study (every 3 weeks) until progression or death (whichever occurs first) up to 374 weeks.
Population: The randomised set. Data only presented for patients with a baseline and at least one post-baseline assessment of ECOG status.
Measure: Number; unit: percentage of participants
Arm/Group | Afatinib 40 Milligram (mg) | Gemcitabine / Cisplatin Chemotherapy
Number analyzed (Participants) | 237 | 110
percentage of participants
  ECOG PS 0 (baseline) 0 (last value) | 11.4 | 21.8
  ECOG PS 1 (baseline) 0 (last value) | 6.8 | 3.6
  ECOG PS 0 (baseline) 1 (last value) | 8.0 | 14.5
  ECOG PS 1 (baseline) 1 (last value) | 67.5 | 51.8
  ECOG PS 0 (baseline) 2 (last value) | 0.4 | 0.0
  ECOG PS 1 (baseline) 2 (last value) | 2.1 | 1.8
  ECOG PS 0 (baseline) 3 (last value) | 0.0 | 0.0
  ECOG PS 1 (baseline) 3 (last value) | 2.1 | 4.5
  ECOG PS 0 (baseline) 4 (last value) | 0.4 | 0.0
  ECOG PS 1 (baseline) 4 (last value) | 1.3 | 1.8

11. Secondary Outcome: Health Related Quality of Life (HRQOL): Time of Deterioration in Coughing
Description: HRQOL as measured by standardised questionnaires (EuropeanOrganisation for Research and Treatment of Cancer (EORTC)) quality of life questionaires (OLQ-C30) and its lung cancer module (QLQ-LC13). Analysis for cough: QLQ-LC13, question 1.
  Time to deterioration was defined as the time from randomisation to a score increase (i.e. worsened) of at least 10 points from baseline (0 to 100 point scale). Patients without deterioration (including those with disease progression) were censored at the date of the last available HRQOL assessment; patients without post-baseline assessments were censored at the date of randomisation. Patients were considered as having deteriorated at the time of death. The median is Kaplan-Meier estimates.
Time Frame: Baseline and throughout the study (every 3 weeks) until progression or death (whichever occurs first) up to 374 weeks.
Population: The randomised set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Afatinib 40 Milligram (mg) | Gemcitabine / Cisplatin Chemotherapy
Number analyzed (Participants) | 242 | 122
months | 31.05 [17.45 to NA] — As only 84 patients (34.7 percent) in Afatinib 40mg deteriorated, the upper limit of the confidence interval was not estimable. | 10.28 [4.63 to NA] — As only 39 patients (32.0 percent) in Gemcitabine / Cisplatin deteriorated, the upper limit of the confidence interval was not estimable.
Statistical Analysis 1: Comparison: Afatinib 40 Milligram (mg) vs Gemcitabine / Cisplatin Chemotherapy; A stratified log-rank test (by the epidermal growth factor receptor (EGFR) mutation category stratification factor used at randomisation) was used to test for the effect of afatinib on HRQOL compared with gemcitabine / cisplatin chemotherapy; Test type: Superiority; p = 0.0001, Log Rank
Statistical Analysis 2: Comparison: Afatinib 40 Milligram (mg) vs Gemcitabine / Cisplatin Chemotherapy; Cox proportional hazard model stratified by EGFR mutation group; Test type: Superiority; Hazard Ratio (HR) = 0.458, 95% CI 2-sided [0.303 to 0.692]

12. Secondary Outcome: Health Related Quality of Life (HRQOL): Time of Deterioration in Dyspnoea
Description: HRQOL as measured by OLQ-C30 and its lung cancer module (QLQ-LC13). Analysis for dyspnoea: composite of QLQ-LC13, questions 3 to 5; individual item from QLQ-C30, question 8.
  Time to deterioration was defined as the time from randomisation to a score increase (i.e. worsened) of at least 10 points from baseline (0 to 100 point scale). Patients without deterioration (including those with disease progression) were censored at the date of the last available HRQOL assessment; patients without post-baseline assessments were censored at the date of randomisation. Patients were considered as having deteriorated at the time of death. The median is Kaplan-Meier estimates.
Time Frame: Baseline and throughout the study (every 3 weeks) until progression or death (whichever occurs first) up to 374 weeks.
Population: The randomised set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Afatinib 40 Milligram (mg) | Gemcitabine / Cisplatin Chemotherapy
Number analyzed (Participants) | 242 | 122
months | 7.66 [4.76 to 11.17] | 1.68 [1.38 to 3.15]
Statistical Analysis 1: Comparison: Afatinib 40 Milligram (mg) vs Gemcitabine / Cisplatin Chemotherapy; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p < 0.0001, Log Rank
Statistical Analysis 2: Comparison: Afatinib 40 Milligram (mg) vs Gemcitabine / Cisplatin Chemotherapy; Cox proportional hazard model stratified by EGFR mutation group; Test type: Superiority; Hazard Ratio (HR) = 0.534, 95% CI 2-sided [0.394 to 0.724]

13. Secondary Outcome: Health Related Quality of Life (HRQOL): Time of Deterioration in Pain
Description: HRQOL as measured by OLQ-C30 and its lung cancer module QLQ-LC13. Analysis for pain: composite of QLQ-C30, questions 9 and 19; individual items from QLQ-LC13, questions 10, 11 and 12.
  Time to deterioration was defined as the time from randomisation to a score increase (i.e. worsened) of at least 10 points from baseline (0 to 100 point scale). Patients without deterioration (including those with disease progression) were censored at the date of the last available HRQOL assessment; patients without post-baseline assessments were censored at the date of randomisation. Patients were considered as having deteriorated at the time of death. The median is Kaplan-Meier estimates.
Time Frame: Baseline and throughout the study (every 3 weeks) until progression or death (whichever occurs first) up to 374 weeks.
Population: The randomised set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Afatinib 40 Milligram (mg) | Gemcitabine / Cisplatin Chemotherapy
Number analyzed (Participants) | 242 | 122
months | 6.93 [4.21 to 10.38] | 3.38 [1.77 to 5.29]
Statistical Analysis 1: Comparison: Afatinib 40 Milligram (mg) vs Gemcitabine / Cisplatin Chemotherapy; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.0220, Log Rank
Statistical Analysis 2: Comparison: Afatinib 40 Milligram (mg) vs Gemcitabine / Cisplatin Chemotherapy; Cox proportional hazard model stratified by EGFR mutation group; Test type: Superiority; Hazard Ratio (HR) = 0.699, 95% CI 2-sided [0.511 to 0.956]

14. Secondary Outcome: Pharmacokinetics of Afatinib at Day 22
Description: Outcome data are the trough plasma concentrations of afatinib at day 22 after multiple daily dosing of 40mg afatinib and after dose escalation to 50mg or dose reduction to 30mg afatinib (no patient dose reduced to 20mg during the Pharmacokinetics (PK) assessment period).
Time Frame: Day 22 (course 2, visit 1)
Population: All patients who had at least 1 afatinib dose and who had at least 1 valid afatinib plasma concentration available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/millilitre (ng/mL)
Groups:
- Afatinib 30mg q.d.: Patients receiving Afatinib 30mg once daily (q.d.) orally after a dose reduction.
- Afatinib 40mg q.d.: Patients receiving Afatinib 40mg once daily (q.d.) orally
- Afatinib 50mg q.d.: Patients receiving Afatinib 50mg once daily (q.d.) orally after a dose escalation.
Arm/Group | Afatinib 30mg q.d. | Afatinib 40mg q.d. | Afatinib 50mg q.d.
Number analyzed (Participants) | 3 | 210 | 0
nanogram/millilitre (ng/mL) | 17.7 (109) | 23.1 (65.1) |

15. Secondary Outcome: Pharmacokinetics of Afatinib at Day 29
Description: Outcome data are the trough plasma concentrations of afatinib at day 29 after multiple daily dosing of 40mg afatinib and after dose escalation to 50mg or dose reduction to 30mg afatinib (no patient dose reduced to 20mg during the PK assessment period).
Time Frame: Day 29 (course 2, visit 2)
Population: All patients who had at least 1 afatinib dose and who had at least 1 valid afatinib plasma concentration available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Afatinib 30mg q.d.: Patients receiving Afatinib 30mg once daily (q.d.) after a dose reduction.
- Afatinib 40mg q.d.: Patients receiving Afatinib 40mg once daily (q.d.)
- Afatinib 50mg q.d.: Patients receiving Afatinib 50mg once daily (q.d.) after a dose escalation.
Arm/Group | Afatinib 30mg q.d. | Afatinib 40mg q.d. | Afatinib 50mg q.d.
Number analyzed (Participants) | 6 | 161 | 34
ng/mL | 19.5 (90.3) | 23.8 (70.6) | 22.8 (60.8)

16. Secondary Outcome: Pharmacokinetics of Afatinib at Day 43
Description: Outcome data are the trough plasma concentrations of afatinib at day 43 after multiple daily dosing of 40mg afatinib and after dose escalation to 50mg or dose reduction to 30mg afatinib (no patient dose reduced to 20mg during the PK assessment period).
Time Frame: Day 43 (course 3, visit 1)
Population: All patients who had at least 1 afatinib dose and who had at least 1 valid afatinib plasma concentration available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Afatinib 30mg q.d. | Afatinib 40mg q.d. | Afatinib 50mg q.d.
Number analyzed (Participants) | 21 | 158 | 35
ng/mL | 21.5 (52.9) | 22.1 (67.4) | 22.9 (62.5)

17. Secondary Outcome: Safety of Afatinib as Indicated by Intensity and Incidence of Adverse Events
Description: Safety of Afatinib as indicated by intensity and incidence of adverse events graded according to the US National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. Presented as the percentage of patients with an Adverse Events during the on-treatment period by highest CTCAE grade.
Time Frame: From first administration of study medication up to 28 days after the last administration of study medication up to 374 weeks.
Population: The treated set (TS) included all randomised patients who were documented to have taken at least 1 dose of study medication (i.e. afatinib or gemcitabine / cisplatin). Patients were allocated according to the treatment actually received.
Measure: Number; unit: percentage of participants
Arm/Group | Afatinib 40 Milligram (mg) | Gemcitabine / Cisplatin Chemotherapy
Number analyzed (Participants) | 239 | 113
percentage of participants
  CTCAE Grade 1 | 13.8 | 8.0
  CTCAE Grade 2 | 36.0 | 29.2
  CTCAE Grade 3 | 39.3 | 38.1
  CTCAE Grade 4 | 4.2 | 21.2
  CTCAE Grade 5 | 6.7 | 2.7

18. Secondary Outcome: Changes in Safety Laboratory Parameters
Description: Outcome data presented are the percentage of patients by worst CTCAE grade (only Grades 2 to 4 presented) on treatment for the following laboratory parameters: Potassium, Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), Creatine and Creatine Kinase.
  For Potassium; only CTCAE grades resulting from hypokalemia (low values) are presented.
Time Frame: as for outcome 17
Population: Treated set (TS) included all randomised patients who were documented to have taken at least 1 dose of study medication. Patients were allocated according to the treatment actually received. Patients with a baseline and at least one on-treatment assessment of the parameter are of interest.
Measure: Number; unit: percentage of participants
Arm/Group | Afatinib 40 Milligram (mg) | Gemcitabine / Cisplatin Chemotherapy
Number analyzed (Participants) | 239 | 113
percentage of participants
  Potassium CTCAE grade 2: number analyzed (Participants) | 235 | 109
  Potassium CTCAE grade 2 | NA — no corresponding rules defined | NA — no corresponding rules defined
  Potassium CTCAE grade 3: number analyzed (Participants) | 235 | 109
  Potassium CTCAE grade 3 | 5.1 | 15.6
  Potassium CTCAE grade 4: number analyzed (Participants) | 235 | 109
  Potassium CTCAE grade 4 | 2.6 | 0.9
  AST CTCAE grade 2: number analyzed (Participants) | 235 | 107
  AST CTCAE grade 2 | 5.1 | 1.9
  AST CTCAE grade 3: number analyzed (Participants) | 235 | 107
  AST CTCAE grade 3 | 1.3 | 1.9
  AST CTCAE grade 4: number analyzed (Participants) | 235 | 107
  AST CTCAE grade 4 | 0.0 | 0.0
  ALT CTCAE grade 2: number analyzed (Participants) | 235 | 108
  ALT CTCAE grade 2 | 8.1 | 5.6
  ALT CTCAE grade 3: number analyzed (Participants) | 235 | 108
  ALT CTCAE grade 3 | 3.4 | 1.9
  ALT CTCAE grade 4: number analyzed (Participants) | 235 | 108
  ALT CTCAE grade 4 | 0.0 | 0.0
  Creatinine CTCAE grade 2: number analyzed (Participants) | 235 | 109
  Creatinine CTCAE grade 2 | 2.1 | 2.8
  Creatinine CTCAE grade 3: number analyzed (Participants) | 235 | 109
  Creatinine CTCAE grade 3 | 0.0 | 0.0
  Creatinine CTCAE grade 4: number analyzed (Participants) | 235 | 109
  Creatinine CTCAE grade 4 | 0.0 | 0.0
  Creatinine Kinase CTCAE grade 2: number analyzed (Participants) | 216 | 104
  Creatinine Kinase CTCAE grade 2 | 3.7 | 1.0
  Creatinine Kinase CTCAE grade 3: number analyzed (Participants) | 216 | 104
  Creatinine Kinase CTCAE grade 3 | 1.9 | 0.0
  Creatinine Kinase CTCAE grade 4: number analyzed (Participants) | 216 | 104
  Creatinine Kinase CTCAE grade 4 | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: From first administration of study medication until 28 days after the last administration of study medication up to 374 weeks
Description: The treated set (TS) included all randomised patients documented to have taken at least 1 dose of study medication. Analysis of Adverse Events (AEs) was based on the concept of treatment-emergent AEs. AEs with onset after the first administration of study drug and within 28 days after the last administration were considered to be on-treatment.
Arm/Group | Afatinib 40 Milligram (mg) | Gemcitabine / Cisplatin Chemotherapy
All-Cause Mortality (participants affected / at risk) | 16/239 | 3/113
Serious Adverse Events (participants affected / at risk) | 40/239 | 12/113
Other Adverse Events (participants affected / at risk) | 236/239 | 112/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 40 Milligram (mg) (N=239) | Gemcitabine / Cisplatin Chemotherapy (N=113)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Cardiac failure (Cardiac disorders) | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Death (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Sudden death (General disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Central nervous system infection (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Meningitis viral (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Embolism (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 40 Milligram (mg) (N=239) | Gemcitabine / Cisplatin Chemotherapy (N=113)
Anaemia (Blood and lymphatic system disorders) | 23 | 31
Leukopenia (Blood and lymphatic system disorders) | 17 | 58
Neutropenia (Blood and lymphatic system disorders) | 13 | 61
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 20
Abdominal discomfort (Gastrointestinal disorders) | 3 | 7
Constipation (Gastrointestinal disorders) | 9 | 31
Diarrhoea (Gastrointestinal disorders) | 212 | 17
Mouth ulceration (Gastrointestinal disorders) | 58 | 2
Nausea (Gastrointestinal disorders) | 28 | 85
Stomatitis (Gastrointestinal disorders) | 52 | 1
Vomiting (Gastrointestinal disorders) | 33 | 91
Asthenia (General disorders) | 17 | 10
Chest pain (General disorders) | 27 | 8
Fatigue (General disorders) | 32 | 35
Mucosal inflammation (General disorders) | 18 | 1
Pain (General disorders) | 12 | 1
Pyrexia (General disorders) | 25 | 12
Nasopharyngitis (Infections and infestations) | 21 | 2
Paronychia (Infections and infestations) | 80 | 0
Upper respiratory tract infection (Infections and infestations) | 17 | 2
Urinary tract infection (Infections and infestations) | 12 | 2
Alanine aminotransferase increased (Investigations) | 58 | 18
Aspartate aminotransferase increased (Investigations) | 47 | 12
Blood creatine phosphokinase increased (Investigations) | 13 | 0
Blood creatinine increased (Investigations) | 11 | 9
Haemoglobin decreased (Investigations) | 6 | 22
Neutrophil count decreased (Investigations) | 2 | 29
Platelet count decreased (Investigations) | 4 | 11
Weight decreased (Investigations) | 33 | 6
White blood cell count decreased (Investigations) | 5 | 27
Decreased appetite (Metabolism and nutrition disorders) | 38 | 47
Hypocalcaemia (Metabolism and nutrition disorders) | 5 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 28 | 26
Hyponatraemia (Metabolism and nutrition disorders) | 7 | 14
Hypoproteinaemia (Metabolism and nutrition disorders) | 14 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 31 | 9
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 18 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 26 | 4
Dizziness (Nervous system disorders) | 22 | 9
Headache (Nervous system disorders) | 30 | 8
Insomnia (Psychiatric disorders) | 13 | 15
Proteinuria (Renal and urinary disorders) | 10 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 47 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 38 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 18 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 17 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 7 | 11
Dry skin (Skin and subcutaneous tissue disorders) | 14 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 16 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 27 | 0
Rash (Skin and subcutaneous tissue disorders) | 175 | 10
Skin fissures (Skin and subcutaneous tissue disorders) | 18 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2013-10-16): https://cdn.clinicaltrials.gov/large-docs/93/NCT01121393/Prot_000.pdf
  • Statistical Analysis Plan (2012-12-05): https://cdn.clinicaltrials.gov/large-docs/93/NCT01121393/SAP_001.pdf